CLINICAL TRIAL: NCT05287074
Title: The Significance of a Timely Food Allergy Diagnosis and Optimal Surveillance of Nutritional Status in Children
Status: Enrolling by invitation | Type: Observational
Sponsor: Vilnius University (Other)
Responsible Party: Sponsor
Other Study IDs: MAMS2018
Record Dates: First submitted 2021-07-14; First posted 2022-03-18 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2021-07

CONDITIONS: Food Allergy in Children; Food Allergy in Infants
Keywords: Food allergy; Milk; Egg
MeSH Terms: conditions — Food Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to gain more knowledge on the nutritional and immunological aspects of allergy to milk and eggs in children.

DETAILED DESCRIPTION:
Food allergy in children is an emerging problem in many countries. Milk and eggs are important sources of nutrition in childhood. Restricting these products in children's diets can affect the quality of child's life and nutrition, which is paramount to good physical and mental child development during this vulnerable period of life. The aim of this study is to gain more knowledge on the nutritional and immunological aspects of immunoglobulin E (IgE) mediated allergy to milk and eggs in children. In this study we will analyze parent perceived child's quality of life, factual nutrition (assessed by 3-day food diaries), food allergy self efficacy measure for parents, parent perceived quality of life will be assessed using Food Allergy Quality of Life Questionnaire - Parent Form, anthropometric measures of children (height and weight), serum nutritional markers (vitamin D, calcium, magnesium, iron and phosphorous), sensitization tests (specific Immunoglobulin E (sIgE) to milk and egg and their components) as well as markers of allergic inflammation (interleukin 10, 13, 17, 25 and 33, eosinophil count and serum Immunoglobulin E). Food allergy will be confirmed by an oral food challenge (OFC), variables will be compared between different OFC outcomes (sensitized-allergic/sensitized-non-allergic).

ELIGIBILITY:
Inclusion Criteria:

* Subjects from 6 months to 12 years of age and their parents / guardians.
* Subjects with suspected or confirmed allergy to chicken's egg and/or cow's milk. Suspected food allergy is defined as sensitization to a food that has not been consumed recently (in the last 3 months) without symptoms or sensitization to a food that has never been consumed. A confirmed food allergy is defined as a food allergy that has previously been confirmed by a positive result of an oral food challenge.
* Legal guardians of the subject are capable to sign a written informed consent form.

Exclusion Criteria:

* Subjects to whom food allergies are unlikely (who have recently eaten a suspected food without symptoms or who have not eaten food recently but have never had symptoms and are not sensitized).
* Subjects to whom an oral food challenge is contraindicated.
* Subjects with comorbid chronic diseases affecting the child 's nutrition and growth.
* Legal guardians of the subject do not wish to participate in the study or are unable to sign a written consent form.

Ages: 6 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Subjects from 6 months to 12 years of age with suspected or confirmed allergy to chicken's egg and/or cow's milk, referred for an oral food challenge with milk or egg will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the daily food intake of children following egg and/or milk elimination diets. | Within one month of enrolment.
  Dietary intake will be assessed by a 3-day food diary, the nutrient intake will be analyzed using national food composition database and a nutritional analysis software.
Antropometric measurements - Z-scores | Within one day of enrolment.
  Anthropometric measurements (weight and height) will be recorded and evaluated as Z-scores using the WHO ANTHRO program and WHO ANTHRO Plus Software.

SECONDARY OUTCOMES:
Evaluation of parental confidence in managing food allergy. | Within one month of enrollment
  Parental confidence will be assessed using Food Allergy Self-Efficacy Scale for Parents (FASE-P), (scale of 0 to 100).
Evaluation of the parent perceived quality of life of children following egg and/or milk elimination diets. | Within one month of enrollment
  Parent perceived quality of life will be assessed using Food Allergy Quality of Life Questionnaire - Parent Form (FAQLQ-PF), (scale of 0 to 6).

OTHER OUTCOMES:
Prick to Prick test with cow's milk mean value. | Within one month of enrollment
  Prick to Prick test with cow's milk mean value.
Prick to Prick test with hen's egg mean value. | Within one month of enrollment
  Prick to Prick test with hen's egg mean value.
Measurement of serum total IgE. | Within one month of enrollment
  Measurement of serum total IgE.
Measurement of serum eosinophils. | Within one month of enrollment
  Measurement of serum eosinophils
Measurement of serum specific IgE to milk extract. | Within one month of enrollment
  Measurement of serum specific IgE to milk extract.
Measurement of serum specific IgE to egg extract. | Within one month of enrollment
  Measurement of serum specific IgE to egg extract.
Measurement of serum specific IgE to casein. | Within one month of enrollment
  Measurement of serum specific IgE to casein.
Measurement of serum specific IgE to betalactoglobulin. | Within one month of enrollment
  Measurement of serum specific IgE to betalactoglobulin.
Measurement of serum specific IgE to ovomucoid. | Within one month of enrollment
  Measurement of serum specific IgE to ovomucoid.
Measurement of serum specific IgE to ovalbumin. | Within one month of enrollment
  Measurement of serum specific IgE to ovalbumin.
Laboratory measurement of vitamin D concentration. | Within one month of enrollment
  Laboratory measurement of vitamin D concentration.
Laboratory measurement of serum calcium concentration. | Within one month of enrollment
  Laboratory measurement of serum calcium concentration.
Laboratory measurement of serum phosphorus concentration. | Within one month of enrollment
  Laboratory measurement of serum phosphorus concentration.
Laboratory measurement of serum iron concentration. | Within one month of enrollment
  Laboratory measurement of serum iron concentration.
Laboratory measurement of serum magnesium concentration. | Within one month of enrollment
  Laboratory measurement of serum magnesium concentration.
Laboratory measurement of serum interleukin 25. | Within one month of enrollment
  Laboratory measurement of serum interleukin 25.
Laboratory measurement of serum interleukin 33. | Within one month of enrollment
  Laboratory measurement of serum interleukin 33.
Laboratory measurement of serum interleukin 17. | Within one month of enrollment
  Laboratory measurement of serum interleukin 17.
Laboratory measurement of serum interleukin 13. | Within one month of enrollment
  Laboratory measurement of serum interleukin 13.
Laboratory measurement of serum interleukin 10. | Within one month of enrollment
  Laboratory measurement of serum interleukin 10.

CONTACTS AND LOCATIONS:
Overall Officials: Ieva Adomaite, MD, Principal Investigator — Vilnius University Faculty of Medicine
Locations (1):
- Vilnius University Hospital Santaros Clinics, Vilnius, Lithuania

IPD SHARING:
Plan to Share IPD: No